CLINICAL TRIAL: NCT00005974
Title: A Phase II Study of Flavopiridol (HMR 1275; NSC 649890) in Patients With Previously Untreated Metastatic or Locally Advanced Soft Tissue Sarcoma
Brief Title: Flavopiridol in Treating Patients With Recurrent, Locally Advanced, or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I136; CAN-NCIC-IND136 (Other: PDQ); NCI-NCIC-136 (Other: NCI); CDR0000067961 (Other: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2004-05-03 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: alvocidib — Flavopiridol 50 mg/m2 IV over 1 hour daily x 3 days every 3 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of flavopiridol in treating patients who have recurrent, locally advanced, or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of flavopiridol in terms of response rate in patients with previously untreated metastatic or locally advanced soft tissue sarcoma. II. Determine the toxicity of this regimen in these patients. III. Determine the time to progression, early progression rate, and response duration in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive flavopiridol IV over 1 hour daily on days 1-3. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed at 4 weeks and then every 3 months until disease progression or death.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study over 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed previously untreated metastatic or locally advanced soft tissue sarcoma not amenable to standard curative therapies Measurable disease At least 20 mm by conventional techniques OR At least 10 mm by spiral CT scan Bone lesions are not considered measurable Must have measurable disease outside irradiated area unless evidence of progression or new lesions inside irradiated area No carcinosarcoma, Kaposi's sarcoma, soft tissue Ewing's sarcoma, or embryonal rhabdomyosarcoma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST no greater than 2.5 times ULN Renal: Creatinine no greater than ULN Cardiovascular: If history of cardiac disease, cardiac ejection function greater than 50% No clinically significant cardiac symptomatology Pulmonary: If history of symptomatic pulmonary disease, FEV1, FVC, and TLC greater than 60% predicted and DLCO greater than 50% predicted No clinically significant pulmonary symptomatology Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent serious disease

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior stem cell transplantation Chemotherapy: No prior chemotherapy for metastatic or locally advanced disease No prior high dose chemotherapy and stem cell transplantation Prior adjuvant chemotherapy allowed At least 6 months since prior chemotherapy No other concurrent cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No more than 25% of functioning bone marrow irradiated No concurrent radiotherapy to sole site of measurable disease Surgery: At least 4 weeks since prior major surgery Other: No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-07-04 (Actual); Primary Completion 2002-11-07 (Actual); Study Completion 2008-09-22 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2 years
  To assess the efficacy (response rate) of flavopiridol given as an N infusion daily x 3 days every 3 weeks in the patients with untreated, metastatic or locally advanced soft tissue sarcoma.

SECONDARY OUTCOMES:
Toxicity | 2 years
  To assess the toxicity of flavopiridol in patients with untreated, metastatic or locally advanced soft tissue sarcoma, as well as time to progression and early progression rate (PD within first 6 weeks), and, if responses are observed, response duration

CONTACTS AND LOCATIONS:
Overall Officials: Donald G. Morris, MD, PhD, FRCPC, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (61):
- St. Mary's/Duluth Clinic Health System, Duluth, Minnesota, United States
- Canada (60):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - Burnaby Hospital Regional Cancer Centre, Burnaby, British Columbia
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - Capital Health Region (Endeavor Clinical Research), Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton and Disrict Urology Association, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Male Health Centre/CMX Research Inc., Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Centre Universitaire de Sante de l'Estrie - Site Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Lions Gate Hospital, North Vancouver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morris DG, Bramwell VH, Turcotte R, Figueredo AT, Blackstein ME, Verma S, Matthews S, Eisenhauer EA. A Phase II Study of Flavopiridol in Patients With Previously Untreated Advanced Soft Tissue Sarcoma. Sarcoma. 2006;2006:64374. doi: 10.1155/SRCM/2006/64374. PMID 17251659